CLINICAL TRIAL: NCT01004939
Title: Retrospektive Studie zu Patientinnen, Die pränatal, Perinatal Oder Postnatal Prophylaktisch Oder Therapeutisch Mit Fondaparinux Behandelt Wurden
Brief Title: Retrospective Study of Patients Who Were Treated With Fondaparinux Pre-, Peri- and/or Postpartum for Prophylaxis or Treatment of Venous Thromboembolism
Acronym: FondaPPP
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Other Study IDs: 112937
Record Dates: First submitted 2009-10-01; First posted 2009-10-30 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-07

CONDITIONS: Thromboembolism; Venous Thromboembolism
Keywords: prophylaxis; venous thromboembolism; postpartum; fondaparinux; pregnancy
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism | interventions — Fondaparinux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fondaparinux prescribed subjects: fondaparinux prescribed subjets
  Interventions: Drug: fondaparinux

INTERVENTIONS:
Drug: fondaparinux — fondaparinux

SUMMARY:
The objective of this retrospective study is to gather information about how fondaparinux is used pre-, peri- and/or postpartum for both the prophylaxis and treatment of venous thromboembolism (VTE) in order to fill an information gap concerning the off-label use of fondaparinux during pregnancy.

DETAILED DESCRIPTION:
During pregnancy there is a generally enhanced risk to develop venous thromboembolism (VTE). Although such events are rare they may lead to serious risks for the mothers´ and children´s health. Compared with non-pregnant women, pregnant women have an about five-fold risk to develop VTE.

Due to their characteristic spectrum of side effects and the generally long duration of exposure in pregnancy the preferred anticoagulants may produce potentially dangerous side effects, as bleedings, heparin-induced thrombocytopenia (HIT), allergic reactions, osteoporosis, or congenital anomalies.

Today, low-molecular weight heparins (LMWH) are the preferred agents for anticoagulation in pregnancy. Compared with unfractioned heparins (UFH) LMWHs have the advantages of a lower bleeding risk, a lower rate of allergic reactions and HIT, a more predictable response and a longer half-life that makes dosing more convenient (od or bid).

Still, there is a considerable proportion of pregnancies where heparin intolerance (allergic reactions or HIT) that make it inevitable to change to another anticoagulant.

On the one hand, fondaparinux has repeatedly been reported successful in the VTE prophylaxis of pregnancies where allergic reactions on heparins, or heparinoids, had occurred. Additionally, a considerable amount of oral reports have reached GSK about an additional number of successful cases in the past.

On the other hand, we have no systematic and overall view about how many pregnancies have already been treated for which reasons, and how successful they were. Due to an increase of certain risk factors, as obesity or the growing age of mothers at childbirth with the associated need for anticoagulation, we expect an increased number of cases where alternative anticoagulation to heparins may be needed.

There are a number of potential advantages of fondaparinux over heparins, such as a once daily application, no dose adjustment needed to body weight and no monitoring of thrombocytes, a lower potential for causing intolerance reactions and no risk for HIT.

The objective of this retrospective study is to gather information about how fondaparinux is used pre-, peri- and/or postpartum for both the prophylaxis and treatment of VTE in order to fill an information gap concerning the off-label use of fondaparinux during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated with fondaparinux pre-, peri- and/or postpartum for more than 7 days for VTE prophylaxis or treatment, especially those with a history of abortion, and/or stillbirth, VTE, severe fetal and maternal complications during pregnancy, severe inherited or acquired thrombophilias, long-term anticoagulation (e. g. patients with mechanical heart valves) and/or intolerance to heparins or heparinoids or heparin-induced thrombocytopenia (HIT)

Exclusion Criteria:

* Patients who were treated with fondaparinux for less than 7 days
* Patient who were treated with fondaparinux only postpartum

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who received a prophylaxis against venous thromboembolism because of an elevated thromboembolic risk and who were therefore treated in a haemostaseological centre.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Germany (7):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin

REFERENCES:
- [Derived] Dempfle CE, Koscielny J, Lindhoff-Last E, Linnemann B, Bux-Gewehr I, Kappert G, Scholz U, Kropff S, Eberle S, Bramlage P, Heinken A. Fondaparinux Pre-, Peri-, and/or Postpartum for the Prophylaxis/Treatment of Venous Thromboembolism (FondaPPP). Clin Appl Thromb Hemost. 2021 Jan-Dec;27:10760296211014575. doi: 10.1177/10760296211014575. PMID 33942675

RESULTS

PARTICIPANT FLOW:
Groups:
- Fondaparinux: Retrospective systematic documentation of female participants treated with Fondaparinux during pregnancy and/or postpartum. The potential prophylactic dose was 1.5 or 2.5 milligrams (mg); the standard prophylactic dose was 2.5 mg. The potential therapeutic dose was 5, 7.5, or 10 mg. Higher than recommended doses could have been administered off label.
Period: Overall Study
Arm/Group | Fondaparinux
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Age Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms (kg)/meters squared (m^2)] — BMI is calculated as body weight in kilograms (kg) divided by body height in meters squared (m^2)
  kilograms (kg)/meters squared (m^2) | 26.5 (6.2)
Number of participants with the indicated anamnestic thromboembolisms [Number; unit: participants] — Known anamnestic (experienced in the past) arterial and venous thromboembolisms, important dispositional risk factors, are reported. A thromboembolism is a clot in the blood that forms and blocks a blood vessel.
  participants
    None | 79
    Arterial only | 0
    Venous only | 39
    Both arterial and venous | 2
Number of participants with known thrombophilia [Number; unit: participants] — Thrombophilic defects, important dispositional risk factors, are reported. It is possible for a participant to have multiple responses. Thrombophilia is a genetic disorder of blood coagulation that increases the risk of thrombosis.
  participants
    None | 20
    Protein C deficiency | 5
    Protein S deficiency | 10
    Antithrombin deficiency | 2
    Factor V Leiden mutation heterozygous | 13
    Factor V Leiden mutation homozygous | 0
    Prothrombin mutation heterozygous | 13
    Prothombin mutation homozygous | 0
    Antiphospholipid syndrome | 15
    Persistant factor VIII increase | 4
    Factor VII activating protease (FSAP) | 6
    Factor VII C46T | 18
    Other | 46
Number of participants with the indicated risk factors for venous thromboembolism [Number; unit: participants] — It is possible for a participant to have more than one of the indicated risk factors.
  participants
    None | 75
    Previous oral contraception | 11
    Hormonotherapy in in-vitro fertilization | 10
    Other supportive gynaecological treatments | 8
    Malignant underlying disease | 3
    Adiposity (BMI>=30) | 12
    Smoking | 11
    Alcohol | 1
    Drug abuse | 1
    Chronic inflammatory disease | 3
    Serious systemic infection | 3
    Immobilization | 5
    Diabetes mellitus | 2
    Hypercholesteremia | 3
    Hypertonia | 5
    Other | 5
Number of participants with the indicated number of former pregnancies [Number; unit: participants]
  Missing | 1
  0 | 35
  1 | 43
  2 | 19
  3 | 15
  4 | 3
  5 | 2
  6 | 1
  10 | 1
Number of participants with the indicated type of former birth [Number; unit: participants] — It is possible for a participant to have more than one type of former birth. It is possible for a participant to have multiple responses.
  participants
    Missing data | 59
    All former births | 61
    Still births | 6
    Live births | 56
    Healthy children | 51
    Children with abnormalities | 1
Number of participants who indicated that they did or did not have former abortions [Number; unit: participants] — Participants were asked to respond "Yes" or "No" to the question: "Did you have former abortions." Only those participants who reported a former pregnancy responded to this question.
  participants
    Total | 85
    Yes | 32
    No | 51
    Missing data | 2
Number of participants with the indicated number of former abortions [Number; unit: participants] — Data were collected from only those participants who gave a response of "Yes" to the question of "Did you have former abortions."
  participants
    Total | 51
    1 | 27
    2 | 16
    3 | 2
    4 | 2
    6 | 1
    Missing data | 3
Number of participants undergoing either prophylaxis or therapy [Number; unit: participants] — The number of participants receiving either antithrombotic prophylaxis (designed and used to prevent a disease from occurring) or therapy of acute venous thromboembolism was measured. It is possible for a participant to have multiple responses.
  participants
    Prophylaxis | 111
    Therapy | 11
Number of participants receiving the indicated type of prophylactic treatment [Number; unit: participants] — A prophylactic treatment is one that is designed and used to prevent a disease from occurring. Prophylaxis for thromboembolic risk is treatment for dispositional thromboembolic risk factors. It is possible for one participant to undergo multiple types of prophylactic treatment.
  participants
    Prophylaxis: thromboembolic risk | 99
    Prophylaxis: surgery | 5
    Prophylaxis: internal medicine | 31
Number of participants receiving therapeutic treatment for the given indications [Number; unit: participants] — It is possible for one participant to undergo multiple types of therapeutic treatment for multiple indications.
  participants
    Data missing | 1
    Therapy: deep vein thrombosis | 7
    Therapy: pulmonary embolism | 3
    Peripheral arterial disease | 0
    Acute coronary syndrome | 0
    Alternative anticoagulation at atrial fibrilation | 0
    Alternative anticoagulation at heart valve | 1
Number of participants receiving thromboembolic prophylaxis for the given indications [Number; unit: participants] — It is possible for one participant to undergo multiple types of treatment for multiple indications. VTE, venous thromboembolis.
  participants
    Thrombophilia | 82
    VTE in anamnesis | 33
    Women with >=2 risk factors | 9
    Long-time anticoagulation with oral anticoagulants | 4
    Antiphospholipid syndrome | 14
    Antithrombine deficiency | 3
    Acute VTE during pregnancy | 1
Number of participants with thrombophilia accompanied by venous thromboembolism (VTE) in anamnesis [Number; unit: participants] — Thrombophilia is a genetic disorder of blood coagulation that increases the risk of thrombosis.
  participants
    Total | 82
    Missing | 2
    Without VTE in anamnesis | 58
    With VTE in anamnesis | 22
Number of participants who did and did not receive UFH [Number; unit: participants] — Unfractionated heparin (UFH) is an anticoagulant.
  participants
    Did not receive UFH | 117
    Received UFH | 3
Duration of UFH administration [Median (Full Range); unit: days] | 32 [7 to 102]
Number of participants with the indicated reason for the end of UFH administration [Number; unit: participants] — It is possible for one participant to have multiple responses.
  participants
    End of thromboembolism prophylaxis/therapy | 1
    Change to another antithrombotic agent | 0
    Thrombocytopenia | 0
    Allergy to heparin | 2
Number of participants receiving the indicated type of low-molecular-weight heparin (LMWH) [Number; unit: participants] — It is possible for one participant to have multiple responses.
  participants
    Total | 120
    Missing | 45
    Enoxaparin | 28
    Nadroparin | 21
    Dalteparin | 35
    Certoparin | 1
    Tinzaparin | 0
    Reviparin | 0
Duration of LMWH administration [Median (Full Range); unit: days] | 54 [4 to 1205]
Number of participants with the indicated reason for the end of LMWH administration [Number; unit: participants] — It is possible for one participant to have multiple responses.
  participants
    Total | 120
    Missing | 44
    End of thromboembolism prophylaxis/therapy | 3
    Change to another antithrombotic agent | 44
    Thrombocytopenia | 7
    Allergy to heparin | 39
    Other | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Fondaparinux in the Indicated Therapy Intervals
Description: The prenatal interval is defined as the interval of time until 3 days before birth. The perinatal interval is defined as the interval of time from 2 days before birth to one day after birth. The postnatal interval is defined as the interval of time beginning 2 days after birth.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010
Measure: Number; unit: participants
Groups:
- Fondaparinux: Retrospective systematic documentation of female patients treated with Fondaparinux during pregnancy and/or postpartum. The potential prophylactic dose was 1.5 or 2.5 milligrams (mg); the standard prophylactic dose was 2.5 mg. The potential therapeutic dose was 5, 7.5, or 10 mg. Higher than recommended doses could have been administered off label.
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Prenatal only | 6
  Perinatal only | 0
  Postnatal only | 1
  Prenatal and Perinatal | 3
  Perinatal and Postnatal | 1
  Prenatal and Postnatal | 2
  Prenatal, Perinatal, and Postnatal | 97
  Unknown | 10

2. Primary Outcome: Number of Participants With the Indicated Reason for Change to Fondaparinux
Description: It was possible for a participant to have changed to fondaparinux for multiple reasons.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Heparin-induced thrombocytopenia (HIT) | 12
  Allergy to heparin | 50
  Other intolerances | 3
  Lack of compliance | 3
  Fix dose | 0
  No monitoring of thrombocyte count necessary | 16
  Medical decision because of other reasons | 42
  Other reasons | 47

3. Primary Outcome: Number of Participants Administered the Indicated Dose of Fondaparinux Per Day
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Dose missing | 2
  2.5 milligrams (mg) | 94
  5 mg | 16
  5 mg until delivery, followed by 2.5 mg | 1
  7.5 mg | 3
  10 mg | 4

4. Primary Outcome: Duration of Fondaparinux Administration
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=101 participants with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 101
days | 131 [2 to 1392]

5. Primary Outcome: Duration of Prenatal Fondaparinux Administration
Description: The prenatal interval is defined as the interval of time until 3 days before birth.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=99 participants with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 99
days | 130 [5 to 468]

6. Primary Outcome: Duration of Postnatal Fondaparinux Administration
Description: The postnatal interval is defined as the interval of time beginning 2 days after birth.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=90 participants with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 90
days | 23 [11 to 41]

7. Primary Outcome: Number of Participants for Whom Fondaparinux Administration Was Interrupted for Birth
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Missing data | 9
  Not interrupted | 20
  Interrupted | 91

8. Primary Outcome: Number of Hours Before Birth That the Last Fondaparinux Dose Was Administered
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=45 participants with non-missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fondaparinux
Number analyzed (Participants) | 45
hours | 34.6 (10.8)

9. Primary Outcome: Number of Hours After Birth at Which Fondaparinux Administration Was Restarted
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=86 participants with non-missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fondaparinux
Number analyzed (Participants) | 86
hours | 11.3 (5.2)

10. Primary Outcome: Number of Participants With the Indicated Reason for the End of Fondaparinux Administration
Description: It is possible that a participant stopped receiving Fondaparinux for multiple reasons.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Missing data | 18
  End of thromboembolism prophylaxis/therapy | 94
  Change to another antithrombotic agent | 6
  Thrombocytopenia (HIT II) | 0
  Allergic reaction | 0
  Other reasons | 5

11. Primary Outcome: Number of Participants With the Indicated Outcome of Pregnancy by Type of Birth
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Missing data | 11
  Spontaneous | 71
  Induced | 3
  Caesarian section | 34
  Induced/Caesarian section | 1

12. Primary Outcome: Number of Participants With the Indicated Type of Conception/Fertilization
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Missing | 2
  Normal conception | 107
  Induced pregnancy with normal conception | 1
  In-vitro fertilization | 10

13. Primary Outcome: Number of Participants Who Delivered a Single Child Versus Twins
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Single child | 116
  Twins | 4

14. Primary Outcome: Mean Weight of Newborn
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Newborns of pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. A total of 124 newborns were born to 120 women; 4 women bore twins. n=63 newborns with non-missing data.
Measure: Mean (Standard Deviation); unit: grams
Units Other Than Participants: newborns
Groups:
- Fondaparinux: Retrospective systematic documentation of female patients treated with Fondaparinux during pregnancy and/or postpartum. The potential prophylactic dose was 1.5 or 2.5 milligrams (mg); the standard prophylactic dose was 2.5 mg. The potential therapeutic dose was 5, 7.5, or 10 mg. Higher than recommended doses could have been administered off label. Data were collected from newborns delivered by participants who received Fondaparinux during pregnancy and/or postpartum.
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Number analyzed (newborns) | 63
grams | 3042 (662.6)

15. Primary Outcome: Mean Height of Newborn
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Newborns of pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. A total of 124 newborns were born to 120 women; 4 women bore twins. n=37 newborns with non-missing data.
Measure: Mean (Standard Deviation); unit: centimeters
Units Other Than Participants: newborns
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Number analyzed (newborns) | 37
centimeters | 49.6 (3.8)

16. Primary Outcome: Mean Head Circumference of Newborn
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Newborns of pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. A total of 124 newborns were born to 120 women; 4 women bore twins. n=27 newborns with non-missing data.
Measure: Mean (Standard Deviation); unit: centimeters
Units Other Than Participants: newborns
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Number analyzed (newborns) | 27
centimeters | 34 (2.2)

17. Primary Outcome: Mean APGAR Score at 1, 5, and 10 Minutes After Birth
Description: APGAR is a test performed by a doctor, midwife, or nurse at 1 and 5 minutes after birth. The 1-minute score determines how well the baby tolerated the birthing process; the 5-minute score assesses how well the newborn is adapting to the new environment. The health care provider examines the baby's breathing effort, heart rate, muscle tone, reflexes, and skin color. Each category is scored with 0 (worst score), 1, or 2 (best score), depending on the observed condition. The rating is based on a total score of 1-10, with 10 suggesting the healthiest infant.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Newborns of pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. A total of 124 newborns were born to 120 women; 4 women bore twins. n=26 (1 min) or n=27 (5 and 10 min) newborns with non-missing data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: newborns
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Number analyzed (newborns) | 27
scores on a scale
  after 1 min, n=26 | 8.6 (0.9)
  after 5 min, n=27 | 9.1 (0.7)
  after 10 min, n=27 | 9.6 (0.5)

18. Primary Outcome: Number of Newborns Who Had a "Healthy" Postnatal Classification
Description: A "healthy" documentation was based on the investigators' individual assessment.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Newborns of pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. A total of 124 newborns were born to 120 women; 4 women bore twins.
Measure: Number; unit: newborns
Units Other Than Participants: newborns
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Number analyzed (newborns) | 124
newborns
  Missing data | 10
  Healthy | 110
  Not healthy | 4

19. Primary Outcome: Number of Newborns With Abnormalities
Description: No formal definition for abnormalities was predetermined; documentation was based on the investigators' individual assessment.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Newborns of pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010
Measure: Number; unit: newborns
Units Other Than Participants: newborns
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
Number analyzed (newborns) | 124
newborns
  Missing data | 10
  No abnormalities | 114

20. Secondary Outcome: Number of Participants Hospitalized Because of Thromboembolic Treatment
Description: Thromboembolic treatment is a defined as prophylaxis for an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  Not hospitalized | 102
  Hospitalized | 18

21. Secondary Outcome: Duration of All Hospitalizations Under UFH, LMWH, and Fondaparinux Administration
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=9 participants with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 9
days | 5 [2 to 28]

22. Secondary Outcome: Duration of Hospitalizations Before, During, and After Fondaparinux Administration
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=3 participants (before Fondaparinux), n=5 participants (during Fondaparinux), and n=1 participant (after Fondaparinux) with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 5
days
  Before Fondaparinux, n=3 | 10 [2 to 28]
  During Fondaparinux, n=5 | 5 [2 to 10]
  After Fondaparinux, n=1 | 2 [2 to 2]

23. Secondary Outcome: Number of Participants With Complications Under UFH/LMWH Therapy
Description: A complication is defined as any thromoemolism, bleeding, skin change, HIT, amputation, or other complication (as indicated by investigator).
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  Missing data | 40
  No complications | 31
  Complications | 49

24. Secondary Outcome: Number of Participants With Thromboembolisms Under UFH/LMWH Therapy
Description: Any sign of thromboembolism as indicated by investigator was measured.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No thromboembolism or missing data | 118
  Thromboembolisms | 2

25. Secondary Outcome: Number of Participants With Bleedings Under UFH/LMWH Therapy
Description: No formal definition for bleeding was predetermined; documentation was based on the investigators' individual assessment.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No bleeding or missing data | 118
  Bleeding | 2

26. Secondary Outcome: Number of Participants With Skin Changes Under UFH/LMWH Therapy
Description: No formal definition for skin change was predetermined; documentation was based on the investigators' individual assessment.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No skin changes or missing data | 80
  Skin changes | 40

27. Secondary Outcome: Duration From Start of UFH/LMWH Therapy to Skin Change
Description: as for outcome 26
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=27 participants with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 27
days | 42 [3 to 134]

28. Secondary Outcome: Number of Participants Who Exhibited Observed Skin Changes and Also Had Erythema Associated With the Skin Changes Under UFH/LMWH Therapy
Description: Erythema is defined as inflammation of the skin, associated with reddening, and is a frequent side effect of heparins.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. Only participants exhibiting skin changes are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 40
participants
  Total | 40
  No erythema or missing data | 4
  Erythema | 36

29. Secondary Outcome: Number of Participants Who Exhibited Observed Skin Changes and Also Had Skin Necrosis Associated With the Skin Changes Under UFH/LMWH Therapy
Description: Skin necrosis is defined as the dying off of skin area because of allergic reaction. Skin necrosis is a severe side effect of heparins.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 40
participants
  Total | 40
  No skin necrosis or missing data | 32
  Skin necrosis | 8

30. Secondary Outcome: Number of Participants With Heparin-induced Thrombocytopenia (HIT II) Under UFH/LMWH Therapy
Description: HIT II is characterized as a sudden decrease of thrombocyte count because of allergic response on heparin/platelet factor 4 (PF-4) complexes and is a severe and potentially fatal side effect of heparins. Usually, HIT occurs between Day 5 and Day 14 of exposure to UFH or LMWH.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No HIT II or missing data | 111
  HIT II | 9

31. Secondary Outcome: Duration From Start of UFH/LMWH Therapy to HIT
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010; n=8 participants with non-missing data.
Measure: Median (Full Range); unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 8
days | 27.5 [3 to 576]

32. Secondary Outcome: Number of Participants With and Without Complications Under Fondaparinux Therapy
Description: A complication is defined as any thromoemolism, bleeding, skin change, HIT, amputation, death, or other complication (as indicated by investigator).
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No complications or missing data | 111
  Complications | 9

33. Secondary Outcome: Number of Participants With Thromboembolisms Under Fondaparinux Therapy
Description: Any sign of thromboembolism as indicated by investigator was measured.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  Either missing data or no thromboembolisms | 120

34. Secondary Outcome: Number of Participants With Bleedings Under Fondaparinux Therapy
Description: as for outcome 25
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No bleedings or missing data | 118
  Bleedings | 2

35. Secondary Outcome: Number of Participants With Skin Changes Under Fondaparinux Therapy
Description: as for outcome 26
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No skin changes or missing data | 120

36. Secondary Outcome: Number of Participants With Heparin-induced Thrombocytopenia (HIT II) Under Fondaparinux Therapy
Description: The participant with HIT II was pretreated with LMWH; however, the serious adverse event of HIT II was documented after the participant switched to Fondaparinux treatment.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fondaparinux
Number analyzed (Participants) | 120
participants
  Total | 120
  No HIT II or missing data | 119
  HIT II | 1

37. Secondary Outcome: Duration From Start of Fondaparinux Therapy to HIT
Description: For the 1 participant who developed HIT after receiving Fondaparinux, the number of days from start of therapy to HIT is presented.
Time Frame: 4 months (all cases occurred between 2004 and 2010)
Population: Pregnant women who received prophylaxis because of an elevated thromboembolic risk or therapeutic treatment of acute thromboembolism between the years of 2004 and 2010. Only one participant developed HIT after receiving Fondaparinux; thus, rather than presenting median data, data are presented as the number of days from start of therapy to HIT.
Measure: Number; unit: days
Arm/Group | Fondaparinux
Number analyzed (Participants) | 1
days | 15

ADVERSE EVENTS:
Groups:
- Fondaparinux - Mother: Events reported for mothers receiving Fondaparinux
- Fondaparinux - Child: Events reported for children (including 4 twins) born to mothers receiving Fondaparinux
Arm/Group | Fondaparinux - Mother | Fondaparinux - Child
Serious Adverse Events (participants affected / at risk) | 9/120 | 1/124
Other Adverse Events (participants affected / at risk) | 6/120 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux - Mother (N=120) | Fondaparinux - Child (N=124)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Heparin-induced thrombocytopenia (General disorders) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Trisomy 18 (Congenital, familial and genetic disorders) | 0 | 1
Transaminases increased (Investigations) | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux - Mother (N=120) | Fondaparinux - Child (N=124)
Drug hypersensitivity (Immune system disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.